CLINICAL TRIAL: NCT01170637
Title: Bioequivalence of a Fixed Dose Combination Tablet Containing 200 mg Ibuprofen and 30 mg Pseudoephedrine-HCl Compared to RhinAdvil® (200 mg Ibuprofen and 30 mg Pseudoephedrine-HCl) as a Fixed Dose Combination Tablet Administered in Healthy Male and Female Volunteers (Open-label, Randomised, Single Dose, Two-way Crossover, Phase I Trial).
Brief Title: Bioequivalence of a Fixed Dose Combination Tablet Containing 200 mg Ibuprofen and 30 mg Pseudoephedrine-HCl Compared to RhinAdvil(R)(200 mg Ibuprofen and 30 mg Pseudoephedrine-HCl) as a Fixed Dose Combination Tablet Administered in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1024.7; 2010-019052-45 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-07-26; First posted 2010-07-27 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Healthy
MeSH Terms: interventions — Ibuprofen; Acetaminophen

ARMS (4):
- Ibuprofen 200 mg (Active Comparator): Oral administration as a fixed dose combination tablet (RhinAdvil(R))
  Interventions: Drug: Ibuprofen
- Pseudoephedrine-HCl 30 mg (Active Comparator): Oral administration as a fixed dose combination tablet (RhinAdvil(R))
  Interventions: Drug: Pseudoephedrine-HCl
- Ibuprofen 200 mg BI (Active Comparator): Oral administration as a fixed dose combination tablet (BI product)
  Interventions: Drug: Ibuprofen
- Pseudoephedrine-HCl 30 mg BI (Active Comparator): Oral administration as a fixed dose combination tablet (BI product)
  Interventions: Drug: Pseudoephedrine-HCl

INTERVENTIONS:
Drug: Ibuprofen — 200 mg oral administration (RhinAdvil(R))
  Arms: Ibuprofen 200 mg
Drug: Ibuprofen — 200 mg oral administration (BI product)
  Arms: Ibuprofen 200 mg BI
Drug: Pseudoephedrine-HCl — 30 mg oral administration (BI product)
  Arms: Pseudoephedrine-HCl 30 mg
Drug: Pseudoephedrine-HCl — 30 mg oral administration (RhinAdvil(R))
  Arms: Pseudoephedrine-HCl 30 mg BI

SUMMARY:
The objective of the current study is to demonstrate bioequivalence of a fixed dose combination tablet containing ibuprofen 200 mg and pseudoephedrine-HCl 30 mg (Test) and RhinAdvil® (Reference) a fixed dose combination tablet containing ibuprofen 200 mg and pseudoephedrine-HCl 30 mg following orally administration.

ELIGIBILITY:
Inclusion criteria

1. Healthy males and females according to the following criteria:

   Based upon a complete medical history, including physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead electrocardiogram (ECG), clinical laboratory tests
2. Age 21 to 50 years
3. BMI 18.5 to 29.9 kg/m2
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion criteria

1. Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Any relevant Gastrointestinal (e.g. ulcera, hernia, bleedings and spasm), hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Any relevant surgery of the gastrointestinal tract (except appendectomy)
5. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
6. History of relevant orthostatic hypotension, fainting spells or blackouts
7. Chronic or relevant acute infections
8. History of relevant allergy or hypersensitivity (including allergy to drug or its excipients) as judged clinically relevant by the investigator
9. Intake of drugs with a long half-life (>24 hours) within at least 1 month or less than 10 half-lives of the respective drug prior to first drug administration
10. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to randomisation
11. Participation in another trial with an investigational drug within 2 months prior to administration or during the trial
12. Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
13. Inability to refrain from smoking on trial days as judged by the investigator
14. Alcohol abuse (average consumption of more than 20 g/day in females and 30 g/day in males)
15. Drug abuse
16. Blood donation (more than 100 mL within four weeks prior to administration of the trial drug in this study)
17. Excessive physical activities within 1 week prior to randomisation or during the trial
18. Any laboratory value outside the reference range that is of clinical relevance
19. Inability to comply with dietary regimen of the study centre
20. Unwilling to avoid excessive sunlight exposure
21. Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval within 10 days prior to administration or during the trial, and CYP2C8 substrates such as amiodarone, amodiaquine, paclitaxel, rosiglitazone, pioglitazone and repaglinide or CYP2C9 such as warfarin, tolbutamide, phenytoin, losartan, acenocoumarol within 1 month or six half lives (whichever is greater)
22. A marked baseline prolongation of the QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
23. A history of additional risk factors for torsade de pointes (e.g., heart failure, hypokalaemia, family history of Long QT Syndrome)

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2010-07; Primary Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of last quantifiable time point) | 1 month
Cmax (maximum measured concentration of the analyte in plasma) | 1 month

SECONDARY OUTCOMES:
AUC0-* (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) (*=infinity) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1024.7.1 Boehringer Ingelheim Investigational Site, Ingelheim, Germany